CLINICAL TRIAL: NCT00859755
Title: A Safety Study of ARRY-403 in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Array BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: ARRAY-403-101
Record Dates: First submitted 2009-03-06; First posted 2009-03-11 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ARRY-403

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- ARRY-403 (Experimental)
  Interventions: Drug: ARRY-403, glucokinase activator; oral
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; oral

INTERVENTIONS:
Drug: ARRY-403, glucokinase activator; oral — single dose, escalating
  Arms: ARRY-403
Drug: Placebo; oral — matching placebo
  Arms: Placebo

SUMMARY:
This is a Phase 1 study, involving a 1-day dosing period, designed to test the safety of investigational study drug ARRY-403 in patients with Type 2 diabetes. Approximately 36 patients from the US will be enrolled in this study.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female with willingness and ability to use protocol-specified methods of contraception, except females of nonchildbearing potential.
* Diagnosis of Type 2 diabetes less than 5 years prior to study start.
* HbA1c ≥ 6.5% and ≤ 10%.
* BMI ≥ 25 and ≤ 40.0 kg/m2.
* Additional criteria exist.

Key Exclusion Criteria:

* Recent history (i.e., less than 6 months) or concomitant/ongoing clinically significant hematologic, renal, pulmonary, gastrointestinal, hepatic, psychiatric, neurologic, dermatologic, or allergic disease (including drug allergies that are clinically significant and not remote, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Significant cardiac disease, myocardial infarction within 6 months of study start, unstable angina, congestive heart failure, known arrhythmias of ventricular etiology, unexplained syncope or syncope/seizures related to arrhythmia.
* History of gastric surgery, vagotomy, bowel resection, or any surgical procedure that might interfere with gastrointestinal motility, pH, or absorption.
* Active infectious diseases including hepatitis B, hepatitis C, or human immunodeficiency virus (HIV). Past history and inactive hepatitis B and C, as confirmed by serological testing, are allowed.
* A positive test for drugs or alcohol.
* Women who are pregnant or breastfeeding.
* Donation or loss of ≥ 550 mL of blood (including plasmapheresis) or receipt of a transfusion of any blood product within 8 weeks prior to first dose of study drug.
* Additional criteria exist.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-03; Primary Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Characterize the safety profile of the study drug in terms of adverse events, clinical laboratory tests, vital signs and electrocardiograms. | Duration of study
Characterize the pharmacokinetics (PK) of the study drug and metabolites in terms of plasma concentrations. | Day 1, Day 2

SECONDARY OUTCOMES:
Characterize the pharmacodynamic (PD) activity of the study drug on biomarkers. | Day 1, Day 2
Assess the ability of the study drug to improve glucose tolerance as determined by blood glucose monitoring during a standardized meal challenge. | Day 1, Day 2
Assess the excretion of the study drug and metabolites in urine following dosing. | Day 1, Day 2

CONTACTS AND LOCATIONS:
Locations (1):
- Profil Institute for Clinical Research, Inc., Chula Vista, California, United States